CLINICAL TRIAL: NCT01157377
Title: Safety and Efficacy Study of AGN-214868 in Patients With Idiopathic Overactive Bladder and Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214868-004
Record Dates: First submitted 2010-07-01; First posted 2010-07-07 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- AGN-214868 total dose 500 ng (Experimental): AGN-214868 injected into the bladder for total dose of 500 ng on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 total dose 1000 ng (Experimental): AGN-214868 injected into the bladder for total dose of 1000 ng on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 total dose 2000 ng (Experimental): AGN-214868 injected into the bladder for total dose of 2000 ng on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 total dose 6000 ng (Experimental): AGN-214868 injected into the bladder for total dose of 6000 ng on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 total dose 18000 ng (Experimental): AGN-214868 injected into the bladder for total dose of 18000 ng on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 total dose 60000 ng (Experimental): AGN-214868 injected into the bladder for total dose of 60000 ng on Day 1.
  Interventions: Drug: AGN-214868
- Placebo to AGN-214868 (Placebo Comparator): Placebo to AGN-214868 injected into the bladder on Day 1.
  Interventions: Drug: AGN-214868 placebo

INTERVENTIONS:
Drug: AGN-214868 — AGN-214868 injected into the bladder.
  Arms: AGN-214868 total dose 1000 ng; AGN-214868 total dose 18000 ng; AGN-214868 total dose 2000 ng; AGN-214868 total dose 500 ng; AGN-214868 total dose 6000 ng; AGN-214868 total dose 60000 ng
Drug: AGN-214868 placebo — AGN-214868 placebo injected into the bladder.
  Arms: Placebo to AGN-214868

SUMMARY:
This study will evaluate the safety and efficacy of AGN-214868 in patients with idiopathic overactive bladder (IOAB) and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be of nonreproductive potential
* If male, must agree to use acceptable contraception
* Symptoms of overactive bladder with urinary urgency incontinence
* Inadequate response or limiting side effects with anticholinergics for the treatment of OAB

Exclusion Criteria:

* Overactive bladder caused by neurological condition (eg, spinal cord injury, multiple sclerosis)
* History of bladder surgery
* Treatment with botulinum toxin therapy of any serotype for any non-urological condition within the prior 12 weeks
* Previous treatment with botulinum toxin therapy of any serotype for any urological condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Richmond, Virginia, United States
- Lyon, France
- Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 160 patients were enrolled, 3 patients did not receive treatment and 1 patient received an incorrect dose. 156 patients were included in the Safety Population.
Period: Overall Study
Arm/Group | AGN-214868 Total Dose 500 ng | AGN-214868 Total Dose 1000 ng | AGN-214868 Total Dose 2000 ng | AGN-214868 Total Dose 6000 ng | AGN-214868 Total Dose 18000 ng | AGN-214868 Total Dose 60000 ng | Placebo to AGN-214868
Started | 23 | 23 | 27 | 15 | 20 | 19 | 29
Completed | 21 | 20 | 26 | 14 | 18 | 16 | 27
Not Completed | 2 | 3 | 1 | 1 | 2 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Personal Reasons | 2 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other Miscellaneous Reasons | 0 | 2 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on the Safety Population that included all participants who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-214868 Total Dose 500 ng | AGN-214868 Total Dose 1000 ng | AGN-214868 Total Dose 2000 ng | AGN-214868 Total Dose 6000 ng | AGN-214868 Total Dose 18000 ng | AGN-214868 Total Dose 60000 ng | Placebo to AGN-214868 | Total
Number analyzed (Participants) | 23 | 23 | 27 | 15 | 20 | 19 | 29 | 156
Age, Customized [Number; unit: Participants]
  < 40 years | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 4
  40-64 years | 16 | 15 | 14 | 9 | 13 | 10 | 16 | 93
  >=65 years | 6 | 7 | 12 | 6 | 7 | 9 | 12 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 23 | 14 | 19 | 18 | 27 | 144
  Male | 0 | 3 | 4 | 1 | 1 | 1 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Daily Average Number of Micturition (Urination) Episodes
Description: The average number of urinary episodes (urination into the toilet) was recorded by a patient bladder diary during 3 consecutive days in the week prior to Baseline and Week 12. A negative change from Baseline indicated improvement (fewer urinary episodes).
Time Frame: Baseline, Week 12
Population: Modified Intent-to-treat population included all randomized participants who received study medication and had post-baseline data available for micturition episodes.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | AGN-214868 Total Dose 500 ng | AGN-214868 Total Dose 1000 ng | AGN-214868 Total Dose 2000 ng | AGN-214868 Total Dose 6000 ng | AGN-214868 Total Dose 18000 ng | AGN-214868 Total Dose 60000 ng | Placebo to AGN-214868
Number analyzed (Participants) | 22 | 23 | 27 | 15 | 19 | 19 | 29
Episodes
  Baseline | 13.7 (4.98) | 12.2 (4.08) | 11.0 (3.44) | 10.6 (2.27) | 11.7 (3.90) | 11.6 (3.23) | 11.0 (2.48)
  Change from Baseline at Week 12 | -2.6 (6.38) | -2.1 (2.45) | -1.3 (4.26) | -0.9 (2.40) | -1.7 (3.90) | -2.7 (2.62) | -1.9 (2.18)

ADVERSE EVENTS:
Arm/Group | AGN-214868 Total Dose 500 ng | AGN-214868 Total Dose 1000 ng | AGN-214868 Total Dose 2000 ng | AGN-214868 Total Dose 6000 ng | AGN-214868 Total Dose 18000 ng | AGN-214868 Total Dose 60000 ng | Placebo to AGN-214868
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/23 | 3/27 | 1/15 | 3/20 | 0/19 | 1/29
Other Adverse Events (participants affected / at risk) | 23/23 | 22/23 | 27/27 | 15/15 | 20/20 | 19/19 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AGN-214868 Total Dose 500 ng (N=23) | AGN-214868 Total Dose 1000 ng (N=23) | AGN-214868 Total Dose 2000 ng (N=27) | AGN-214868 Total Dose 6000 ng (N=15) | AGN-214868 Total Dose 18000 ng (N=20) | AGN-214868 Total Dose 60000 ng (N=19) | Placebo to AGN-214868 (N=29)
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0/20 | 0/23 | 1/14 | 0/19 | 0/18 | 0/27
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AGN-214868 Total Dose 500 ng (N=23) | AGN-214868 Total Dose 1000 ng (N=23) | AGN-214868 Total Dose 2000 ng (N=27) | AGN-214868 Total Dose 6000 ng (N=15) | AGN-214868 Total Dose 18000 ng (N=20) | AGN-214868 Total Dose 60000 ng (N=19) | Placebo to AGN-214868 (N=29)
Dysuria (Renal and urinary disorders) | 6 | 5 | 4 | 1 | 3 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 2 | 2 | 0 | 3 | 1
Haematuria (Renal and urinary disorders) | 1 | 2 | 5 | 2 | 4 | 2 | 5
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 1 | 4 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 3 | 0 | 4 | 2 | 3
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 1 | 1 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1/20 | 0/23 | 1/14 | 1/19 | 1/18 | 1/27
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device failure (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydroureter (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0/20 | 0/23 | 1/14 | 0/19 | 0/18 | 0/27
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 4 | 2 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.